CLINICAL TRIAL: NCT03220035
Title: NCI-COG Pediatric MATCH (Molecular Analysis for Therapy Choice)- Phase 2 Subprotocol of Vemurafenib in Patients With Tumors Harboring BRAF V600 Mutations
Brief Title: Vemurafenib in Treating Patients With Relapsed or Refractory Advanced Solid Tumors, Non-Hodgkin Lymphoma, or Histiocytic Disorders With BRAF V600 Mutations (A Pediatric MATCH Treatment Trial)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2017-01244; NCI-2017-01244 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); APEC1621G; APEC1621G (Other: Children's Oncology Group); APEC1621G (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2017-07-17; First posted 2017-07-18 (Actual); Results first posted 2023-09-13 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Advanced Malignant Solid Neoplasm; Ann Arbor Stage III Childhood Non-Hodgkin Lymphoma; Ann Arbor Stage IV Childhood Non-Hodgkin Lymphoma; Ependymoma; Ewing Sarcoma; Hepatoblastoma; Langerhans Cell Histiocytosis; Malignant Germ Cell Tumor; Malignant Glioma; Osteosarcoma; Peripheral Primitive Neuroectodermal Tumor; Recurrent Childhood Central Nervous System Neoplasm; Recurrent Childhood Non-Hodgkin Lymphoma; Recurrent Malignant Solid Neoplasm; Recurrent Neuroblastoma; Refractory Malignant Solid Neoplasm; Refractory Neuroblastoma; Refractory Non-Hodgkin Lymphoma; Refractory Primary Central Nervous System Neoplasm; Rhabdoid Tumor; Rhabdomyosarcoma; Soft Tissue Sarcoma; Wilms Tumor
MeSH Terms: conditions — Ependymoma; Sarcoma, Ewing; Hepatoblastoma; Histiocytosis, Langerhans-Cell; Glioma; Osteosarcoma; Neuroectodermal Tumors, Primitive, Peripheral; Central Nervous System Neoplasms; Neuroblastoma; Lymphoma, Non-Hodgkin; Rhabdoid Tumor; Rhabdomyosarcoma; Sarcoma; Wilms Tumor | interventions — Vemurafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (vemurafenib) (Experimental): Patients receive vemurafenib PO BID on day 1-28. Cycles repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Vemurafenib

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Vemurafenib — Given PO
  Other Names: BRAF (V600E) kinase inhibitor RO5185426; BRAF(V600E) Kinase Inhibitor RO5185426; PLX 4032; PLX-4032; PLX4032; RG 7204; RG-7204; RG7204; RO 5185426; RO-5185426; Zelboraf

SUMMARY:
This phase II Pediatric MATCH trial studies how well vemurafenib works in treating patients with solid tumors, non-Hodgkin lymphoma, or histiocytic disorders with BRAF V600 mutations that have spread to other places in the body (advanced) and have come back (recurrent) or do not respond to treatment (refractory). Vemurafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the objective response rate (ORR; complete response + partial response) in pediatric patients treated with vemurafenib with advanced solid tumors (including central nervous system [CNS] tumors), lymphomas or histiocytic disorders that harbor activating BRAF V600 mutations.

SECONDARY OBJECTIVES:

I. To estimate the progression free survival in pediatric patients treated with vemurafenib with advanced solid tumors (including CNS tumors), lymphomas or histiocytic disorders that harbor activating BRAF V600 mutations.

II. To obtain information about the tolerability of vemurafenib in children with relapsed or refractory cancer.

EXPLORATORY OBJECTIVE:

I. To explore approaches to profiling changes in tumor genomics over time through evaluation of circulating tumor deoxyribonucleic acid (DNA).

OUTLINE:

Patients receive vemurafenib orally (PO) twice daily (BID) on day 1-28. Cycles repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have enrolled onto APEC1621SC and must have been given a treatment assignment to Molecular Analysis for Therapy Choice (MATCH) to APEC1621G based on the presence of a BRAF V600 mutation
* Patients must have a body surface area >= 0.55 m^2 at enrollment; patients < 0.73 m^2 must follow the dosing nomogram; patients >= 0.73 m^2 at enrollment must follow the dosing nomogram
* Patients must have radiographically measurable disease at the time of study enrollment; patients with neuroblastoma who do not have measurable disease but have metaiodobenzylguanidine (MIBG) positive (+) evaluable disease are eligible; measurable disease in patients with CNS involvement is defined as tumor that is measurable in two perpendicular diameters on magnetic resonance imaging (MRI) and visible on more than one slice; Note: The following do not qualify as measurable disease:

  * Malignant fluid collections (e.g., ascites, pleural effusions)
  * Bone marrow infiltration except that detected by MIBG scan for neuroblastoma
  * Lesions only detected by nuclear medicine studies (e.g., bone, gallium or positron emission tomography [PET] scans) except as noted for neuroblastoma
  * Elevated tumor markers in plasma or cerebrospinal fluid (CSF)
  * Previously radiated lesions that have not demonstrated clear progression post radiation
  * Leptomeningeal lesions that do not meet the measurement requirements for Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Karnofsky >= 50% for patients > 16 years of age and Lansky >= 50 for patients =< 16 years of age; Note: Neurologic deficits in patients with CNS tumors must have been stable for at least 7 days prior to study enrollment; patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Patients must have fully recovered from the acute toxic effects of all prior anti-cancer therapy and must meet the following minimum duration from prior anti-cancer directed therapy prior to enrollment; if after the required timeframe, the numerical eligibility criteria are met, e.g. blood count criteria, the patient is considered to have recovered adequately

  * Cytotoxic chemotherapy or other anti-cancer agents known to be myelosuppressive

    * >= 21 days after the last dose of cytotoxic or myelosuppressive chemotherapy (42 days if prior nitrosourea)
  * Anti-cancer agents not known to be myelosuppressive (e.g. not associated with reduced platelet or absolute neutrophil count [ANC] counts): >= 7 days after the last dose of agent
  * Antibodies: >= 21 days must have elapsed from infusion of last dose of antibody, and toxicity related to prior antibody therapy must be recovered to grade =< 1
  * Corticosteroids: If used to modify immune adverse events related to prior therapy, >= 14 days must have elapsed since last dose of corticosteroid
  * Hematopoietic growth factors: >= 14 days after the last dose of a long-acting growth factor (e.g. pegfilgrastim) or 7 days for short-acting growth factor; for growth factors that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur; the duration of this interval must be discussed with the study chair and the study-assigned research coordinator
  * Interleukins, interferons and cytokines (other than hematopoietic growth factors): >= 21 days after the completion of interleukins, interferon or cytokines (other than hematopoietic growth factors)
  * Stem cell Infusions (with or without total-body irradiation [TBI]):

    * Allogeneic (non-autologous) bone marrow or stem cell transplant, or any stem cell infusion including donor lymphocyte infusion (DLI) or boost infusion: >= 84 days after infusion and no evidence of graft versus host disease (GVHD)
    * Autologous stem cell infusion including boost infusion: >= 42 days
  * Cellular therapy: >= 42 days after the completion of any type of cellular therapy (e.g. modified T cells, natural killer [NK] cells, dendritic cells, etc.)
  * Radiation therapy (XRT)/external beam irradiation including protons: >= 14 days after local XRT; >= 150 days after TBI, craniospinal XRT or if radiation to >= 50% of the pelvis; >= 42 days if other substantial bone marrow (BM) radiation; Note: Radiation may not be delivered to "measurable disease" tumor site(s) being used to follow response to subprotocol treatment
  * Radiopharmaceutical therapy (e.g., radiolabeled antibody, iobenguane I-131 [131I-MIBG]): >= 42 days after systemically administered radiopharmaceutical therapy
  * Patients must not have received prior exposure to a BRAF inhibitor (e.g. vemurafenib, dabrafenib or encorafenib)
* For patients with solid tumors without known bone marrow involvement:

  * Peripheral absolute neutrophil count (ANC) >= 1000/mm^3
  * Platelet count >= 100,000/mm^3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment)
* Patients with known bone marrow metastatic disease will be eligible for study provided they meet the blood counts in above criteria (may receive transfusions provided they are not known to be refractory to red cell or platelet transfusions); these patients will not be evaluable for hematologic toxicity
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 ml/min/1.73 m^2 or a serum creatinine based on age/gender as follows:

  * Age: 1 to < 2 years; maximum serum creatinine (mg/dL): male 0.6; female 0.6
  * Age: 2 to < 6 years; maximum serum creatinine (mg/dL): male 0.8; female 0.8
  * Age: 6 to < 10 years; maximum serum creatinine (mg/dL): male 1; female 1
  * Age: 10 to < 13 years; maximum serum creatinine (mg/dL): male 1.2; female 1.2
  * Age: 13 to < 16 years; maximum serum creatinine (mg/dL): male 1.5; female 1.4
  * Age: >= 16 years; maximum serum creatinine (mg/dL): male 1.7; female 1.4
* Bilirubin (sum of conjugated + unconjugated) =< 1.5 x upper limit of normal (ULN) for age
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 135 U/L; (for the purpose of this study, the ULN for SGPT is 45 U/L)
* Serum albumin >= 2 g/dL
* Corrected QT (QTc) interval =< 480 milliseconds; Note: Patients should avoid concomitant medication known or suspected to prolong QTc interval or cause Torsades De Pointes; if possible, alternative agents should be considered; patients who are receiving drugs that prolong the QTc are eligible if the drug is necessary and no alternatives are available
* Patients must be able to swallow intact tablets
* All patients and/or their parents or legally authorized representatives must sign a written informed consent; assent, when appropriate, will be obtained according to institutional guidelines

Exclusion Criteria:

* Pregnant or breast-feeding women will not be entered on this study due to risks of fetal and teratogenic adverse events as seen in animal/human studies; pregnancy tests must be obtained in girls who are post-menarchal; males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method, for the duration of study treatment and for 6 months after the last dose of vemurafenib
* Patients receiving corticosteroids who have not been on a stable or decreasing dose of corticosteroid for at least 7 days prior to enrollment are not eligible; if used to modify immune adverse events related to prior therapy, >= 14 days must have elapsed since last dose of corticosteroid
* Patients who are currently receiving another investigational drug are not eligible
* Patients who are currently receiving other anti-cancer agents are not eligible
* Patients who are receiving cyclosporine, tacrolimus or other agents to prevent graft-versus-host disease post bone marrow transplant are not eligible for this trial
* Patients who are currently receiving drugs that are moderate to strong inducers or inhibitors of CYP3A4 are not eligible; moderate to strong inducers or inhibitors of CYP3A4 should be avoided from 14 days prior to enrollment to the end of the study; Note: CYP3A4 inducing anti-epileptic drugs and dexamethasone for CNS tumors or metastases, on a stable dose, are allowed
* Patients who are currently receiving drugs that are inhibitors or inducers of p-glycoprotein (P-gp) or adenosine triphosphate (ATP)-binding cassette, subfamily G, member 2 (ABCG2 [BCRP]) are not eligible
* Patients with known active cutaneous squamous cell carcinoma (includes keratoacanthoma or mixed keratoacanthoma subtype) are not eligible; patients who have fully excised lesions with dermatologic confirmation of absence of disease are eligible
* Patients with low grade glioma patients (World Health Organization [WHO] grades I and II) are not eligible
* Patients who have an uncontrolled infection are not eligible
* Patients who have received a prior solid organ transplantation are not eligible
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible

Ages: 12 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AeRang Kim, Principal Investigator — Children's Oncology Group
Locations (116):
- United States (114):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Banner Children's at Desert, Mesa, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - UMC Cancer Center / UMC Health System, Lubbock, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Puerto Rico (2):
  - San Jorge Children's Hospital, San Juan
  - University Pediatric Hospital, San Juan

REFERENCES:
- [Derived] Nelson MV, Kim A, Williams PM, Roy-Chowdhuri S, Patton DR, Coffey BD, Reid JM, Piao J, Saguilig L, Alonzo TA, Berg SL, Ramirez NC, Jaju A, Fox E, Weigel BJ, Hawkins DS, Mooney MM, Takebe N, Tricoli JV, Janeway KA, Seibel NL, Parsons DW. Phase II study of vemurafenib in children and young adults with tumors harboring BRAF V600 mutations: NCI-COG pediatric MATCH trial (APEC1621) Arm G. Oncologist. 2024 Aug 5;29(8):723-e1093. doi: 10.1093/oncolo/oyae119. PMID 38873934
- [Derived] Hattinger CM, Patrizio MP, Magagnoli F, Luppi S, Serra M. An update on emerging drugs in osteosarcoma: towards tailored therapies? Expert Opin Emerg Drugs. 2019 Sep;24(3):153-171. doi: 10.1080/14728214.2019.1654455. Epub 2019 Aug 14. PMID 31401903

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Vemurafenib)
Started | 4
Completed | 0
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Protocol Violation | 1
Not completed — Progressive Disease | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Vemurafenib)
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.3 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR will be defined as complete response + partial response and assessed by Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1). Will be calculated as the percent of evaluable patients who are responders, and confidence intervals will be constructed using the Wilson score interval method.
Time Frame: From enrollment to the end of treatment, up to 2 years
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Vemurafenib)
Number analyzed (Participants) | 4
percentage of participants | 25 [5.8 to 64.4]

2. Secondary Outcome: Progress Free Survival (PFS)
Description: PFS will be defined as time from the initiation of protocol treatment to the I of any of the following events: disease progression or disease recurrence or death from any cause. Patients with local calls of disease progression (i.e. calls made by the treating institution), will be counted as having had an event, even if the central review does not declare progression. PFS along with the confidence intervals will be estimated using the Kaplan-Meier method.
Time Frame: From the initiation of protocol treatment to the occurrence of any of the following events: disease progression or disease recurrence or death from any cause, assessed up to 5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Vemurafenib)
Number analyzed (Participants) | 4
percentage of participants | 75 [12.8 to 96.1]

3. Secondary Outcome: Percentage of Patients Experiencing Grade 3 or Higher Adverse Events
Description: Percentage of patients experiencing grade 3 or higher adverse events will be evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. All patients who receive at least one dose of protocol therapy will be considered in the evaluation of toxicity.
Time Frame: From enrollment to 30 days after the end of treatment, up to 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Vemurafenib)
Number analyzed (Participants) | 4
percentage of participants | 75 [19.4 to 99.4]

4. Other Pre Specified Outcome: Changes in Tumor Genomics
Description: Will explore approaches to profiling changes in tumor genomics over time through evaluation of circulating tumor deoxyribonucleic acid. Will be summarized with simple summary statistics and will be descriptive in nature.
Time Frame: Baseline up to 4.5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse Events monitored/assessed from enrollment to 30 days after the end of treatment, up to 2 years. All-Cause Mortality monitored/assessed up to 5 years
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. Ineligible patients are excluded from reporting of adverse events. All-Cause Mortality includes all deaths collected on the study.
Arm/Group | Treatment (Vemurafenib)
All-Cause Mortality (participants affected / at risk) | 1/4
Serious Adverse Events (participants affected / at risk) | 3/4
Other Adverse Events (participants affected / at risk) | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Vemurafenib) (N=4)
Cardiac arrest (Cardiac disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Vemurafenib) (N=4)
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Fever (General disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
White blood cell decreased (Investigations) | 1
Glucose intolerance (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1
Confusion (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-10): https://cdn.clinicaltrials.gov/large-docs/35/NCT03220035/Prot_SAP_000.pdf